CLINICAL TRIAL: NCT07319975
Title: Comparison of the Effects of Semaglutide and Tirzepatide Treatments in Combination With Exercise in Obesity Management
Brief Title: Effect of Semaglutide and Tirzepatide Combined With Exercise in Obesity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Galata University (Other)
Collaborators: Biruni University (Other); Istanbul University (Other)
Responsible Party: Principal Investigator, Safak Yigit, Assistant Professor, Istanbul Galata University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-GLP1-OBESITY
Record Dates: First submitted 2025-12-07; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — semaglutide; Tirzepatide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ARM 1-Semaglutide (Experimental): Drug: Semaglutide
  Interventions: Drug: Semaglutide
- ARM 3-Semaglutide + Exercise (Experimental)
  Interventions: Behavioral: Semaglutide+Exercise
- ARM 4-Tirzepatide + Exercise (Experimental)
  Interventions: Behavioral: Tirzepatide+Exercise
- ARM 2-Tirzepatide (Experimental): Drug: Tirzepatide
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Semaglutide — They will use only semaglutide.
  Arms: ARM 1-Semaglutide
Drug: Tirzepatide — They will use only tirzepatide.
  Arms: ARM 2-Tirzepatide
Behavioral: Tirzepatide+Exercise — This group will engage in exercise and receive tirzepatide therapy."
  Arms: ARM 4-Tirzepatide + Exercise
Behavioral: Semaglutide+Exercise — This group will engage in exercise and receive semaglutide therapy."
  Arms: ARM 3-Semaglutide + Exercise

SUMMARY:
Obesity is a growing global health problem that affects people of all ages. It can lead to serious health issues such as cardiovascular disease, insulin resistance, inflammation, and reduced physical function. New medications, including GLP-1 receptor agonists like semaglutide and dual GLP-1/GIP agonists like tirzepatide, have been shown to help people lose significant weight. However, some of this rapid weight loss may come from a reduction in muscle mass rather than fat. Losing muscle can lower physical performance, impair metabolic health, and increase the risk of developing sarcopenic obesity. This study aims to compare the effects of pharmacological treatment alone with a combined treatment program that includes both medication and exercise in individuals with obesity. The primary objective is to evaluate how these two approaches influence body composition.

The secondary objective is to examine the effects of pharmacological treatment versus combined treatment on cardiometabolic markers, peripheral muscle strength, functional capacity, respiratory function, respiratory muscle performance, and physical activity levels. The study seeks to determine whether adding structured exercise to medication can provide additional health benefits beyond weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 25 and 60 years
* Those with a body mass index (BMI) between 30 and 40 kg/m2 according to the World Health Organization (WHO) classification
* Individuals who volunteered to participate in the study

Exclusion Criteria:

* Individuals with a BMI greater than 40 kg/m2 according to the WHO classification
* Individuals with a Charlson comorbidity index score of 3 or higher
* Uncontrolled arrhythmia, hypertension, heart failure, diabetes, and unstable angina pectoris
* Cooperation impairment, orthopedic, and neurological problems that may interfere with evaluation and treatment
* Individuals with a history of lower extremity injury or surgery in the last six months
* Diagnosed with diabetes and complications such as nephropathy, retinopathy, and neuropathy
* Individuals with concomitant chronic respiratory disease
* Individuals with acute infections
* Individuals with middle ear pathologies (such as tympanic membrane rupture, otitis media)
* Individuals with a history of spontaneous or trauma-related pneumothorax
* Smokers
* Pregnancy
* Individuals with a STOP-bang score of 3 or higher
* Individuals on a structured diet program for weight loss during the study period
* Individuals who have had endoscopic intervention and/or bariatric surgery within the last year

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Body fat-muscle ratios (Body composition) | Three months
  These measurements will be determined by bioelectrical impedance.

SECONDARY OUTCOMES:
Peripheral muscle strength | Three months
  M. Quadriceps muscle strength and hand grip strength measurement will be used to evaluate peripheral muscle strength (kg). Hand-held dynamometer will be used to evaluate quadriceps muscle strength and hand grip strength (kg).
Glucose profile | Three months
  Glucose profile after 12 hours of fasting will be measured. (mg/dL)
Functional capacity | Three months
  Submaximal functional exercise capacity of the participants will be evaluated with the six-minute walk test.
Pulmonary function | Three months
  Spirometric assessment will be performed to determine participants' forced expiratory volume in one second (FEV1). Spirometric assessment will be performed to determine participants' forced vital capacity (FVC).
Respiratory muscle strength | Three months
  Respiratory muscle strength; It will be evaluated with an intraoral pressure measuring device in a sitting position.
Physical activity level | Three months
  Step Count Measurement: Daily step count will be monitored to determine the physical activity level of the participants. Step count will be assessed with a wearable activity monitor, a portable, easy-to-use tool that can measure objectively (Huawei Watch Fit Special Edition). With its six-axis sensor, the device records the user's physical activity style information in its temporary memory throughout the duration of use. Participants will be asked to wear the activity monitor on their left wrist throughout and only remove it during bathing. After one week of use, the data recorded with the wearable activity monitor will be taken.
Incremental load test (Respiratory Muscle Endurance) | Three months
  Respiratory muscle endurance will be evaluated by incremental load test. The incremental load test will be performed using the electronic inspiratory loading device (PowerBreathe®-KHP2).
Lipid Profile | Three months
  Lipid profile after 12 hours of fasting will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No